CLINICAL TRIAL: NCT05034042
Title: A Randomized, Placebo-Controlled, Double-Blind, Phase 2 Study to Select the Optimal Dose(s) of Fezolinetant in Women Suffering From Vasomotor Symptoms (Hot Flashes) Associated With Menopause in Japan
Brief Title: A Study to Find the Best Dose of Fezolinetant to Treat Hot Flashes in Women Going Through Menopause
Acronym: Starlight
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2693-CL-0206; jRCT2031210334 (Registry Identifier: jRCT)
Record Dates: First submitted 2021-09-01; First posted 2021-09-05 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2024-10

CONDITIONS: Hot Flashes
Keywords: Vasomotor Symptoms (Hot Flashes) Associated with Menopause; ESN364; fezolinetant
MeSH Terms: conditions — Hot Flashes | interventions — fezolinetant

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Fezolinetant: low dose (15 mg) (Experimental): Participants will receive low dose of fezolinetant once daily for 12 weeks.
  Interventions: Drug: Fezolinetant
- Fezolinetant: high dose (30 mg) (Experimental): Participants will receive high dose of fezolinetant once daily for 12 weeks.
  Interventions: Drug: Fezolinetant
- Placebo (Placebo Comparator): Participants will receive matching placebo once daily for 12 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Fezolinetant — oral
  Other Names: ESN364
  Arms: Fezolinetant: high dose (30 mg); Fezolinetant: low dose (15 mg)
Drug: Placebo — oral
  Arms: Placebo

SUMMARY:
This study is for menopausal women who have hot flashes. Menopause, a normal part of life, is the time after a woman's last period. Hot flashes often occur during menopause. They can disrupt a woman's daily life. This study will take place in Japan.

This study will provide more information on a potential new treatment, called fezolinetant. The treatments in this study are fezolinetant or a placebo. In this study, a placebo is a dummy treatment that looks like fezolinetant but does not have any medicine in it. The study will compare fezolinetant with the placebo to find the best dose of fezolinetant to reduce the number and severity of hot flashes.

Women that want to take part in the study will be given an electronic handheld device to track their hot flashes. In the last 10 days before their next clinic visit, the women will record information about their hot flashes. Women will be picked for 1 of 3 treatments (lower or higher dose of fezolinetant, or placebo) by chance alone.

Women who take part in the study will take 2 tablets every day for 12 weeks. Treatment will be double-blinded. That means that the women in the study and the study doctors will not know who takes which of the study medicines (lower or higher dose of fezolinetant, or placebo). The women will continue recording information about their hot flashes on the electronic device. They will also use another device to answer questions about how hot flashes affect their daily life.

During the study, the women will visit their study clinic several times for a check-up. This will happen during weeks 2, 4, 8, 12 and 15. At the check-up, they will be asked if they have any medical problems. Other checks will include some blood samples taken for laboratory tests. At some check-ups, the women will have a physical exam, an ECG to check their heart rhythm, and their vital signs checked (pulse rate, temperature and blood pressure). At the first visit and in week 15, women who have a uterus will also have a test called a transvaginal ultrasound. A probe is gently placed inside the vagina. Sound waves will create a picture of the organs in the pelvis. This will allow the study doctor to look more closely at the uterus and surrounding organs.

The last check-up (at week 15) will be 3 weeks after they take their last tablets of study medicine (lower or higher dose of fezolinetant or placebo).

ELIGIBILITY:
Inclusion Criteria:

* Subject has a body mass index ≥ 16 kg/m^2 and ≤ 38 kg/m^2 at screening visit.
* Subject must be seeking treatment or relief for vasomotor symptoms (VMS) associated with menopause and confirmed as menopausal per 1 of the following criteria at the screening visit:

For post-menopausal subjects:

* Spontaneous amenorrhea for ≥ 12 consecutive months
* Spontaneous amenorrhea for ≥ 6 months with biochemical criteria of menopause (follicle-stimulating hormone [FSH] > 40 IU/L); or
* Having had bilateral oophorectomy ≥ 6 weeks prior to the screening visit (with or without hysterectomy)

For peri-menopausal subjects:

* Skipped menstrual period with amenorrhea for ≥ 60 days but < 6 consecutive months with biochemical criteria of peri-menopause (FSH > 25 IU/L); or
* Spontaneous amenorrhea for ≥ 6 months but < 12 consecutive months with biochemical criteria of peri-menopause (FSH > 25 IU/L and ≤ 40 IU/L)

  * Within the 10 days prior to randomization, subject must have a minimum average of 7 mild, moderate and severe hot flashes (VMS) per day.
  * Subject is not pregnant and at least 1 of the following conditions apply:
* Not a woman of childbearing potential (WOCBP)
* WOCBP who agrees to follow the contraceptive guidance from the time of informed consent through at least 21 days after the final study treatment administration

  * Subject must agree not to breastfeed starting at screening and throughout the study period and for 21 days after the final study treatment administration.
  * Subject must not donate ova starting at first dose of investigational product (IP) and throughout the study period and for 21 days after the final study treatment administration.
  * Subject is in good general health as determined on the basis of medical history and general physical examination, including a bimanual clinical pelvic examination and clinical breast examination devoid of relevant clinical findings, performed at the screening visit; hematology and biochemistry parameters, pulse rate and/or blood pressure, and electrocardiogram (ECG) within the reference range for the population studied, or showing no clinically relevant deviations.
  * Subject has documentation of a normal/negative or no clinically significant abnormal findings on breast imaging (obtained at screening or within the prior 12 months of screening). Appropriate documentation includes a written report or an electronic report indicating normal/negative or no clinically significant abnormal findings on breast imaging.
  * Subject is willing to undergo a transvaginal ultrasound (TVU) to evaluate the uterus and ovaries at screening and week 12 (end of treatment), and for subjects who are withdrawn from the study prior to completion, a TVU at the early discontinuation visit. This is not required for subjects who have had a partial (supra-cervical) or full hysterectomy.
  * Subject is willing to undergo endometrial biopsy at any time during the study in the case of uterine bleeding. This is not required for subjects who have had a partial (supra-cervical) or full hysterectomy and for peri-menopausal subjects in case of menstrual bleeding.
  * Subject has documentation of a normal or not clinically significant abnormal Pap test (or equivalent cervical cytology) within the previous 12 months of screening or at screening. This is not required for subjects who have had a full trachelectomy.
  * Subject has a negative urine pregnancy test at screening. Urine pregnancy test is not required for female subjects who are assessed as post-menopausal status.
  * Subject has negative serology panel (i.e. negative hepatitis B surface [HBs] antigen) and negative hepatitis C virus [HCV] antibody) at screening.
  * Subject agrees not to participate in another interventional study while participating in the present study.

Exclusion Criteria:

* Subject uses a prohibited therapy (strong or moderate cytochrome P450 1A2 [CYP1A2] inhibitors, hormone replacement therapy [HRT], hormonal contraceptive or any treatment for VMS [prescription, over the counter, or herbal/Chinese medicine]) or is not willing to wash out and discontinue use of such drugs for the full duration of study conduct or it is not medically appropriate to discontinue such drugs for the duration of the study.
* Subject has known substance abuse or alcohol addiction within 6 months of screening.
* Subject has a history of a malignant tumor except for non-metastatic basal cell carcinoma of the skin.
* Subject has uncontrolled hypertension.
* Subject has a history of severe allergy, hypersensitivity, or intolerance to drugs in general, including the IP and any of its excipients.
* For subjects with a uterus: Subject has an unacceptable result from the TVU assessment at screening, (i.e., full length of endometrial cavity cannot be visualized or presence of a clinically significant abnormal finding).
* Subject has a history of an undiagnosed uterine bleeding within the previous 6 months of screening.
* Subject has a history of seizures or other convulsive disorders.
* Subject has a medical condition or chronic disease (including history of neurological [including cognitive], hepatic, renal, cardiovascular, gastrointestinal, pulmonary [e.g., moderate asthma], endocrine, or gynecological disease) or malignancy that could confound interpretation of the study outcome.
* Subject has active liver disease, jaundice, or elevated liver aminotransferases (alanine aminotransferase [ALT] or aspartate aminotransferase [AST]), elevated total or direct bilirubin, elevated international normalized ratio (INR), or elevated alkaline phosphatase (ALP) at screening. Subject with mildly elevated ALT or AST up to < 1.5 × the upper limit of normal (ULN) can be enrolled if total and direct bilirubin are normal. Subject with mildly elevated ALP (up to < 1.5 × ULN) can be enrolled if cholestatic liver disease is excluded and no cause other than fatty liver is diagnosed. Subject with Gilbert's syndrome with elevated total bilirubin (TBL) may be enrolled as long as direct bilirubin (DBL), hemoglobin and reticulocytes are normal.
* Subject has creatinine > 1.5 × ULN; or estimated glomerular filtration rate (eGFR) using the Modification of Diet in Renal Disease formula ≤ 59 mL/min/1.73 m^2 at screening visit.
* Subject has a previous positive test for the human immunodeficiency virus.
* Subject has a history of suicide attempt or suicidal behavior within the prior to 12 months of study enrollment or has suicidal ideation within the prior to 12 months of study enrollment (a response of "yes" to question 4 or 5 on the suicidal ideation portion of the Columbia Suicide Severity Rating Scale [C-SSRS]), or who is at significant risk to commit suicide at screening and at visit 2.
* Subject has had previous exposure with fezolinetant.
* Subject has received an IP within 28 days or 5 half-lives, whichever is longer, prior to screening.
* Subject is unable or unwilling to complete the study procedures.
* Subject has any condition which makes the subject unsuitable for study participation.
* Subject or relative is the investigator or other site staff directly involved in the conduct of the study.
* Subject is an employee of the sponsor, contract research organizations (CROs) or site management organizations (SMOs).
* Present or previous history of participation in a study of the IP.

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 147 (Actual)
Dates: Start 2021-11-17 (Actual); Primary Completion 2022-11-11 (Actual); Study Completion 2022-12-23 (Actual)

PRIMARY OUTCOMES:
Mean change from baseline in the frequency of mild, moderate and severe vasomotor symptom (VMS) | Baseline and Week 8
  Frequency of mild, moderate or severe VMS events will be calculated as the sum of mild, moderate or severe VMS events per day.

SECONDARY OUTCOMES:
Mean change from baseline in the frequency of mild, moderate and severe VMS | Baseline and up to Week 12
  Frequency of mild, moderate or severe VMS events will be calculated as the sum of mild, moderate or severe VMS events per day.
Number of participants with Adverse Events (AEs) | Up to Week 15
  An AE is any untoward medical occurrence in a subject administered an investigational product (IP), and which does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of IP whether or not considered related to the IP.
Change from baseline in endometrial thickness | Baseline and Week 12
  Endometrial thickness is a measure of how thick the lining of the uterus is. Endometrial thickness will be measured by transvaginal ultrasound (TVU).
Number of participants with laboratory value abnormalities and/or AEs | Up to Week 15
  Number of participants with potentially clinically significant laboratory values.
Number of participants with vital sign abnormalities and/or AEs | Up to Week 15
  Number of participants with potentially clinically significant vital sign values.
Number of participants with electrocardiogram (ECG) abnormalities and/or AEs | Up to Week 12
  Number of participants with potentially clinically significant ECG values.
Number of participants with suicidal ideation and/or behavior as assessed by Columbia-Suicide Severity Rating Scale (C-SSRS) | Up to Week 15
  The Columbia-Suicide Severity Rating Scale (C-SSRS) is a clinician administered assessment tool that evaluates suicidal ideation and behavior. Number of participants that have an affirmative response provided to the 5 items for suicidal ideation (1. Wish to be dead, 2. Non-specific active suicidal thoughts, 3. Active suicidal ideation with any methods (not plan) without intent to act, 4. Active suicidal ideation with some intent to act, without specific plan, 5. Active suicidal ideation with specific plan and intent) and/or to the 5 items for suicidal behavior (1. Preparatory acts or behavior, 2. Aborted attempt, 3. Interrupted attempt, 4. Actual attempt, 5. Completed suicide) will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Inc
Locations (40):
- Japan (40):
  - Juno Vesta Clinic Hatta, Matsudo-shi, Chiba
  - Mori Ladies Clinic, Fukuoka, Fukuoka
  - SANO Women's Clinic, Fukuoka, Fukuoka
  - Japan Organization of Occupational Health and Safety Kyushu Rosai Hospital, Kitakyusyu-shi, Fukuoka
  - Ena Odori Clinic, Sapporo, Hokkaido
  - Kotoni Ladies Clinic, Sapporo, Hokkaido
  - M's Ladies Clinic, Sapporo, Hokkaido
  - Nishikawa Women's Health Clinic, Sapporo, Hokkaido
  - Sapporo Medical Center, NTT East Corporation, Sapporo, Hokkaido
  - Tonan Hospital, Sapporo, Hokkaido
  - Asahi-Clinic, Takamatsu, Kagawa-ken
  - Unoki Clinic, Kagoshima, Kagoshima-ken
  - Yoshinaga Women's Clinic, Kagoshima, Kagoshima-ken
  - Sophia Ladies Clinic, Sagamihara-shi, Kanagawa
  - Tawada Ladies Clinic, Yokohama, Kanagawa
  - Women's Clinic LUNA Yokohama Motomachi, Yokohama, Kanagawa
  - Kyoto City Hospital, Kyoto, Kyoto
  - Chieko Yukika Lady's Clinic, Sendai, Miyagi
  - Social Medical Care Corporation Hosei-kai Marunouchi Hospital, Matsumoto-shi, Nagano
  - Kurashiki Medical Clinic, Kurashiki-shi, Okayama-ken
  - GyNet Medical Corporation Minamimorimachi Ladies' Clinic, Osaka, Osaka
  - Nomura Clinic Namba, Osaka, Osaka
  - jMOG Medical Corporation Tanabe Ladies' Clinic, Takatsuki-shi, Osaka
  - Maruyama Memorial General Hospital, Saitama-shi, Saitama
  - Omi Medical Center, Social Medical Corporation Seikoukai, Kusatsu-shi, Shiga
  - Omihachiman Community Medical Center, Ōmihachiman, Shiga
  - Hamada Hospital, Chiyoda-ku, Tokyo
  - Ginza Yoshida Clinic, Chuo-Ku, Tokyo
  - Medical Corporation Asbo Tokyo Asbo Clinic, Chuo-ku, Tokyo
  - Medical Corp. SEIKOUKAI New Medical Research System Clinic, Hachioji-shi, Tokyo
  - Toranomon Womens Clinic, Minato-ku, Tokyo
  - Yokokura Clinic, Minato-ku, Tokyo
  - Shimamura Memorial Hospital, Nerima-ku, Tokyo
  - Yukawa Women's Clinic, Nishi-Tokyo-shi, Tokyo
  - Seijo Kinoshita Hospital, Setagaya-ku, Tokyo
  - Ikebukuro Clinic, Toshima-ku, Tokyo
  - Ikebukuro Metropolitan Clinic, Toshima-ku, Tokyo
  - Kurobe City Hospital, Kurobe-shi, Toyama
  - Japan Organization of Occupational Health and Safety Toyama Rosai Hospital, Uozu-shi, Toyama
  - Japan Community Healthcare Organization Tokuyama Central Hospital, Shunan-shi, Yamaguchi

IPD SHARING:
Plan to Share IPD: Yes
Access to anonymized individual participant level data collected during the study, in addition to study-related supporting documentation, is planned for studies conducted with approved product indications and formulations, as well as products terminated during development. Studies conducted with product indications or formulations that remain active in development are assessed after study completion to determine if Individual Participant Data can be shared. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Access to participant level data is offered to researchers after publication of the primary manuscript (if applicable) and is available as long as Astellas has legal authority to provide the data.
Access Criteria: Researchers must submit a proposal to conduct a scientifically relevant analysis of the study data. The research proposal is reviewed by an Independent Research Panel. If the proposal is approved, access to the study data is provided in a secure data sharing environment after receipt of a signed Data Sharing Agreement.
URL: https://www.clinicaltrials.astellas.com/transparency/

REFERENCES:
- See also: Link to plain language summary of the study on the Trial Results Summaries website. — https://www.trialsummaries.com/Study/StudyDetails?id=14511&tenant=MT_AST_9011